CLINICAL TRIAL: NCT07047378
Title: Acceptance and Commitment Therapy-Based Training Programme for Reducing Parental Burnout and Improving Emotional and Behavioural Issues in Children: A Pilot Randomised Controlled Trial
Brief Title: ACT-Based Training for Parental Burnout and Child Well-being
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Harmony House (Unknown); Hong Kong Jockey Club (Unknown)
Responsible Party: Principal Investigator, Yuen Yu CHONG, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NTEC-2025-184
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Child Abuse; Parental Burnout
Keywords: Child maltreatment; Acceptance and Commitment Therapy (ACT); Hong Kong; Parental burnout; Psychological flexibility; Feasibility; Acceptability; Child adjustment; Child emotion; Emotional development
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Parallel Assignment; Repeated measures (baseline, post-intervention, and 3-month follow-up) 2-arm randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor(s) is/are blind to the group assignment in this study since it employs single-blind masking. Because of the nature of the intervention, both participants and care providers (e.g., facilitator or therapist) are aware of the assigned condition. To minimize bias in data interpretation, the outcome assessor(s) do/does not have access to participant group assignment information.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT Intervention Group (Experimental): Both ACT Intervention and the Control Group will receive standard services originally provided by Harmony House. For parents allocated to this experimental group, 6 sessions of the ACT-based parenting program, one weekly session, 90 minutes per session. For children allocated to this experimental group, 6 sessions of the child-focused ACT programme, one weekly session, 90 minutes per session.
  Interventions: Behavioral: ACT Intervention Group
- Control Group (Other): Participants allocated to the Control Group will not receive the ACT intervention during the initial 3-month study period but will be offered the intervention afterward as part of a waitlist control design.
  Interventions: Other: control group

INTERVENTIONS:
Behavioral: ACT Intervention Group — For Parent ACT Group, parents will participate in a six-week, group-based ACT program integrated with behavioral parenting training based on positive parenting principles. Each session lasts two hours and includes 65 minutes of ACT-based activities (e.g., experiential exercises, guided imagery, mindfulness, values clarification, metaphors) and 25 minutes of parenting education and/or behavioral skills training.
  For Children ACT Group, children (aged 6-11) will also receive a child-focused ACT intervention to help them manage emotional challenges. Each session lasts two hours and includes 65 minutes of ACT-based activities (e.g., experiential exercises, guided imagery, mindfulness, values clarification, metaphors) and 25 minutes of behavioral skills training.
  Arms: ACT Intervention Group
Other: control group — Participants allocated to the Control Group will not receive the ACT intervention but will continue to receive the standard services originally provided by Harmony House. These services constitute usual care and include initial assessments, individual counselling, group counselling, the provision of community resource information, and referrals. Control group participants will receive these supports as usual. This study will not alter their existing service arrangements in any way, nor will it add to or reduce the support they receive.
  Aside from not participating in the ACT program, the control group's experience will be identical to that of clients receiving regular services. After the intervention group completes the program, the control group will be offered the same course content (i.e., a waitlist intervention arrangement).
  Arms: Control Group

SUMMARY:
The purpose of the proposed randomized controlled trial is to evaluate the feasibility, acceptability, and potential effectiveness of Acceptance and Commitment Therapy (ACT) in reducing parental burnout and improving children's emotional and behavioral adjustment in families in Hong Kong over 3 months after the intervention. The findings will provide valuable and scientific insights to inform better parenting interventions and child protection policies.

DETAILED DESCRIPTION:
Parental burnout is becoming more widely recognized as a serious social issue. It is particularly prevalent among high-stress families like those impacted by child maltreatment or domestic violence. According to prior research, psychological flexibility-a core component of Acceptance and Commitment Therapy (ACT)-is crucial for promoting healthy parent-child relationships and adaptive parenting practices. However, there is still a dearth of empirical evidence supporting ACT-based interventions for reducing parental burnout and improving child adjustment.

The purpose of this study is to investigate how ACT interventions differ in their impact on parents and children in Hong Kong. The specific aims are to evaluate the effectiveness of an ACT-based training program in lowering parental burnout and investigate its influence on children's emotional and behavioral adjustment.

Parents will participate in an ACT-based parenting training program designed to increase psychological flexibility in the ACT intervention group. Aiming at improving psychological flexibility and reducing parental burnout, the training program incorporates mindfulness, values-based parenting, and cognitive defusion strategies. It provides parents with the resources they require to manage stress, regulate emotions, and promote parent-child relationships, which benefits both themselves and their children.

To foster emotional regulation and resilience, children aged 6-11 will also participate in a group-based, child-focused ACT Program designed for their developmental needs. This program incorporates experiential learning exercises, mindfulness activities, and storytelling using picture books to facilitate participation and engagement. These child-focused components seek to reinforce the skills parents have learned while directly supporting child adjustment.

This study aims to examine the feasibility, acceptability, and potential efficacy of a group-based Acceptance and Commitment Therapy (ACT) intervention targeting. The intervention is designed to improve parental psychological flexibility and parenting behaviour, enhance parent- child relationships, and child-related outcomes within a separate sample of parents and children over the 3- month post-intervention. The study will be conducted in collaboration with Harmony Home Limited, leveraging the expertise of paraprofessionals trained in ACT.

ELIGIBILITY:
Inclusion Criteria:

For the Parent ACT Group:

1. Cantonese-speaking Hong Kong residents between the ages of 19 and 65 years.
2. Primary caregivers of a child aged 3 to 11 years.
3. Have been identified by school social workers as being at risk of domestic violence or experiencing emotional distress.

For the Child ACT Group:

1. Cantonese-speaking Hong Kong residents between the ages of 3 and 11 years.
2. Have been identified by school social workers as being at risk of domestic violence or experiencing emotional distress.

For both groups (Shared inclusion criteria):

1. Participants must have sufficient Cantonese language proficiency to understand and communicate during the intervention.
2. Both parents and children must provide informed consent to participate in the study and all related assessments.

Exclusion Criteria:

For the Parent ACT Group:

1. Parents diagnosed with severe mental illnesses.
2. Parents with a developmental disability that interferes with their ability to comprehend the program's content.
3. Parents with cognitive, language, communication, visual, or hearing impairments or disorders that could impede their understanding of the intervention content; or
4. Parents currently participate in other psychosocial, psychoeducational, or parenting interventions.
5. Parents with active substance abuse issues that may interfere with their ability to participate in or benefit from the program.
6. Parents whose children have been diagnosed with psychological or medical conditions.

For the Child ACT Group:

1. Children who have been diagnosed with psychological or medical conditions.

For both groups (Shared Exclusion criteria):

1. Families who are unable or unwilling to commit to attending the six-week sessions or completing follow-up assessments.
2. Families who lack access to transportation or other necessary resources to attend the intervention sessions
3. Parents and children who cannot understand or communicate in the language used in the intervention and assessments (i.e., Cantonese and Chinese).

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Parental Burnout | Change from baseline assessment to immediate and 3 months post-intervention
  The Parental Burnout Assessment (PBA, 23-item, 7-point Likert scale) will be employed to evaluate the level of parental burnout. The Chinese version of PBA has reported good internal consistency (Cronbach's α = >.8), adequate construct validity (.66~.79), and strong convergent validity in Chinese parents.
Children's emotional and behavioral adjustment | Change from baseline assessment to immediate and 3 months post-intervention
  The Strengths and Difficulties Questionnaire (SDQ, 25-item, 3-point Likert scale) will be used to assess children's emotional and behavioral adjustment. The Chinese version of SDQ demonstrates satisfactory internal consistency (Cronbach's α = .45-.90) and good test-retest reliability (coefficients = 0.8 to 0.85).

SECONDARY OUTCOMES:
Parental Psychological flexibility | Change from baseline assessment to immediate and 3 months post-intervention
  Parental Psychological Flexibility Questionnaire (PPFQ, 16-item, 7-point Likert scale) will be employed to measure parents' psychological flexibility. The PPFQ measures psychological flexibility using three subscales: cognitive defusion, committed action, and acceptance. The total and each subscale scores of the Chinese version of PPFQ have demonstrated substantial discriminant and criterion validity and internal consistency (Cronbach's α = .77-.86), and test-retest reliability coefficients ranging from 0.55 to 0.75.
Children's psychological flexibility | Change from baseline assessment to immediate and 3 months post-intervention
  Child and Adolescent Mindfulness Measure (CAMM, 10-item, 5-point Likert scale) will be used to assess children's psychological flexibility through children's self-reports. Grounded in Acceptance and Commitment Therapy (ACT), it measures present-moment awareness and non-judgmental acceptance of thoughts and feelings. The Chinese version of CAMM demonstrates good internal consistency (Cronbach's α = .826) and strong construct validity and acceptable criterion-related validity among Chinese primary school students.
Adaptive parenting behaviors | Change from baseline assessment to immediate and 3 months post-intervention
  Interpersonal Mindfulness in Parenting Scale (IM-P, 31-item, 5-point Likert scale), a parent self-report measure, will be employed to measure adaptive parenting behaviors. The IM-P assesses five dimensions: Listening with Full Attention, Emotional Awareness of Self and Child, Self-Regulation in Parenting, Non-Judgmental Acceptance of Self and Child, and Compassion for Self and Child. The Chinese version of the IM-P was found to have adequate internal consistency (Cronbach's α = 0.85) and has been demonstrated to be a valid measure among Chinese populations.
Parent-Child Relationship Quality | Change from baseline assessment to immediate and 3 months post-intervention
  Child-Parent Relationship Scale-Short Form (CPRS-SF, 15-item, 5-point Likert scale), a parent self-report measure, will be used to assess the quality of the parent- child relationship. The Chinese version of CPRS-SF assesses child-parent relationships across two subscales: conflict and closeness. The internal consistency of the subscales is typically reported as being in the range of 0.70 to 0.90, indicating good reliability.

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - Harmony House Limited, Kwun Tong
  - Chinese University of Hong Kong, Shatin

IPD SHARING:
Plan to Share IPD: No
As participants were not asked to provide consent for sharing their individual data with external researchers, IPD cannot be made available.